CLINICAL TRIAL: NCT02864966
Title: A 24 Hour Occlusive Single Patch Test to Assess, Under Dermatological Control, the Acute Cutaneous Tolerance of Pre Lubricated Kiss Condom on a Panel of Healthy Adult Subjects
Brief Title: A 24 Hour Occlusive Single Patch Test to Assess Acute Tolerance of Pre Lubricated Condom on a Panel of Healthy Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Alba Science Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NPD81401
Record Dates: First submitted 2016-07-28; First posted 2016-08-12 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Safety study; new product; normal healthy skin.
MeSH Terms: interventions — Condoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Other (Other): This is a safety study where a marketed product will be placed on healthy adult skin.
  Interventions: Device: Condom

INTERVENTIONS:
Device: Condom — This study involves testing a condom, however the device will not be used as intended. The device will be destroyed to make the test patches required for this safety study.
  Other Names: Durex

SUMMARY:
This is a 24 hour patch test to determine the acute tolerance of 3 variants of condom on a panel of healthy adult subjects. The patches will be affixed to the back and remain under occlusion for 24 hours. They will then be assessed at 30 minutes and 24 hours post patch removal.

DETAILED DESCRIPTION:
Three test products (plus positive and negative control) will be applied to the back using occlusive tape and will remain on the skin for 24 hours. The patches will be removed after 24 hours and assessed as 30 minutes post patch removal and again at 24 hours post patch removal. Each test site will be scored for erythema and oedema by a dermatologist.

The primary endpoint for this Clinical Investigation is the irritation of the test products according to the Cutaneous Irritancy Index value. The test products success criteria is to be graded as 'non-irritant' and this should be confirmed by the study dermatologist.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to give written informed consent and from whom written informed consent has been obtained
* Generally healthy male or female subjects between the ages of 18 and 70 years inclusive.
* Subjects assessed by the dermatologist as having normal/healthy skin.
* Subjects with skin Phototype I to IV skin.
* Subjects who have been exposed to Natural Rubber Latex through condom use with no allergic reaction being raised
* Subjects, who are able to understand the study, co-operate with the study procedures (including no swimming during the study period) and are able to attend all study assessments.

Exclusion Criteria:

* Female subjects who are pregnant, lactating or have given birth within the previous 3 months or are planning to be pregnant during the study.
* Female subjects of childbearing potential who, for the duration of the study, are either unwilling or unable to take adequate contraceptive precautions or are unwilling to be sexually abstinent.
* Subjects with previous experience of intolerance or allergic reactions to any components of the test products including latex and lubricants.
* Subjects with either form of diabetes.
* Subjects with an active skin disorder or a significant history of skin disorders (e.g. psoriasis, eczema, vitiligo, pityriasis versicolor, acne) which in the opinion of the Principle Investigator or dermatologist may affect the test results
* Subjects whose skin has been excessively exposed to the sun or to UV rays during the previous month in the opinion of the Investigator.
* Subjects who are suffering from chronic asthma, a malfunction of the lymphatic system or an autoimmune deficiency diseases (e.g. lupus, thyroiditis).
* Subjects with very easily irritated/sensitive skin in the opinion of the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the irritation of the test products according to the Cutaneous Irritancy Index value. The test products are expected to be graded as 'non-irritant' as confirmed by a dermatologist. | 24 hours
  Acute tolerance study to test the safety of a new condom on healthy adult skin.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Reynolds, Principal Investigator — Alba Science Ltd
Locations (1):
- Alba Science Ltd, Edinburgh, United Kingdom